CLINICAL TRIAL: NCT01743859
Title: Sequential Treatment With Azacitidine and Lenalidomide for Relapsed and Refractory Patients With Acute Myeloid Leukemia
Brief Title: Azacitidine and Lenalidomide for Relapsed and Refractory Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-1283.cc; NCI-2012-03191 (Other: National Cancer Institute)
Record Dates: First submitted 2012-11-16; First posted 2012-12-06 (Estimated); Results first posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: Myeloid; Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — Azacitidine; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Azacitidine + Lenalidomide + Off Therapy (Experimental): Patients will receive 7 days of azacitidine followed by 3 weeks of lenalidomide. They will then have 2 weeks off therapy, for a maximum of 12 cycles.
  Interventions: Drug: Azacitidine; Drug: Lenalidomide; Other: Off Therapy

INTERVENTIONS:
Drug: Azacitidine — Enrolled patients will receive 75 mg/m2 of azacitidine subcutaneously (SC) or intravenously (IV) on days 1-7 alone.
  Other Names: Vidaza (TM)
Drug: Lenalidomide — Beginning on day 8, patients will receive 50 mg of lenalidomide PO, and will take this daily from day 8 through 28.
  Other Names: Revlimid (TM)
Other: Off Therapy — 2 weeks off therapy, then begin sequence again for 12 weeks.

SUMMARY:
The primary objective of this study is to determine the complete remission/complete remission with incomplete recovery of blood counts (CR/CRi) rate for relapsed and refractory acute myeloid leukemia (AML) and high-risk myelodysplastic syndrome (MDS) patients.

DETAILED DESCRIPTION:
AML patients with relapsed and refractory disease have very poor outcomes. Sequential azacitidine and lenalidomide was recently shown by the PI of this study to be well-tolerated and effective in elderly, treatment naïve AML patients. Observations from this study and others that have piloted this combination have suggested that patients who received and failed prior treatments may also respond to this regimen. Therefore, the sequential combination of azacitidine with lenalidomide could potentially improve outcomes for relapsed and refractory AML patients by providing them with a treatment option that is tolerable and potentially clinically synergistic. To determine the efficacy of this combination in this population, we will pilot this phase 2 study.

ELIGIBILITY:
Inclusion Criteria:

* • World Health Organization (WHO)-confirmed AML, other than Acute Promyelocytic Leukemia (APL)

  * Age >18 years
  * White blood cell count (WBC) at initiation of treatment ≤ 10,000/L

    o If WBC is > 10,000/L patients may be started on an appropriate dose of hydroxyurea (to be determined by the investigators), until WBC < 10,000/L, at which time the hydroxyurea will be discontinued for 12 hours prior to enrollment
  * Relapsed or refractory (resistant) disease, as defined by standard criteria21:

    * Relapsed: Bone marrow blasts ≥5%; reappearance of blasts in the blood; development of extramedullary disease
    * Refractory (resistant): Failure to achieve Complete Remission (CR) or complete remission with incomplete recovery of blood counts (CRi) in patients who survive ≥7 days following completion of initial treatment, with evidence of persistent leukemia by blood and/or bone marrow examination
  * Failure of at least one prior therapy
  * Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (See Appendix D: ECOG Performance Status Scale)
  * Life expectancy > 2 months
  * All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist® (RevAssist is a restricted distribution program for receiving lenalidomide)
  * Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 million International Units per milliliter (mIU/mL) 10 - 14 days prior to study enrollment and again within 24 hours of prescribing lenalidomide (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin two acceptable methods of birth control, one highly effective method and one additional effective method at the same time, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. See Appendix F: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods
  * Willing and able to understand and voluntarily sign a written informed consent
  * Able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

* • Known or suspected hypersensitivity to azacitidine or mannitol

  * Patients with advanced malignant hepatic tumors.
  * Treatment less than four weeks prior to enrollment with other experimental therapies or antineoplastic agents, with the exception of hydroxyurea
  * Inability to swallow or absorb drug
  * Prior treatment with lenalidomide for AML
  * Active opportunistic infection or treatment for opportunistic infection within four weeks of first day of study drug dosing
  * New York Heart Association Class III or IV heart failure
  * Unstable angina pectoris
  * Significant uncontrolled cardiac arrhythmias
  * Uncontrolled psychiatric illness that would limit compliance with requirements
  * Known Human immunodeficiency virus (HIV) infection
  * Graft vs. host disease ≥ grade 2
  * Relapse after allogeneic stem cell transplantation prior to post-transplant day 30
  * Pregnant or breast feeding females; lactating females must agree not to breast feed while taking lenalidomide
  * Other medical or psychiatric illness or organ dysfunction or laboratory abnormality which in the opinion of the investigator would compromise the patient's safety or interfere with data interpretation
  * Laboratory abnormalities:

    * Either creatinine >2.0 mg/dL or creatinine clearance <30 mL/min
    * Total bilirubin > 2 x institutional upper limit of normal (ULN) (unless documented Gilbert's syndrome)
    * Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) > 3 x institutional ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-12-06 (Actual); Primary Completion 2016-04-27 (Actual); Study Completion 2016-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pollyea, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Cancer Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Azacitidine + Lenalidomide + Off Therapy: Patients will receive 75 mg/m2 of azacitidine subcutaneously (SC) or intravenously (IV) on days 1-7 alone. Afterwards beginning on Day 8 patients will receive 50 mg of lenalidomide PO, and will take this daily from day 8 through 28. They will then enter a 2 week observation period where they will be monitored and assessed.
Period: Overall Study
Arm/Group | Azacitidine + Lenalidomide + Off Therapy
Started | 37
Completed | 28
Not Completed | 9

BASELINE CHARACTERISTICS:
Population: Relapsed and refractory AML patients who received azacitidine and lenalidomide
Arm/Group | Azacitidine + Lenalidomide + Off Therapy
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 6
  >=65 years | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Remission or Complete Remission With Incomplete Recovery Blood Counts
Description: Change in baseline to end of study. To be assessed by standard criteria based on bone marrow examination. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Interim assessment after 18 patients (estimated 2 years) and full assessment after 37 patients (estimated 3-4 years)
Population: Relapsed/refractory AML patients who received azacitidine and lenalidomide
Measure: Number; unit: percentage of participants
Arm/Group | Azacitidine + Lenalidomide + Off Therapy
Number analyzed (Participants) | 37
percentage of participants | 11

2. Primary Outcome: Overall Response Rate
Description: Change in baseline to end of study. To be assessed by standard criteria based on bone marrow examination
Time Frame: Planned assessment after enrollment of all 37 patients (estimated 3-4 years)
Population: relapsed/refractory patients who received azacitidine and lenaldiomide
Measure: Number; unit: percentage of participants
Arm/Group | Azacitidine + Lenalidomide + Off Therapy
Number analyzed (Participants) | 37
percentage of participants | 52

3. Secondary Outcome: Response or Remission Duration
Description: Change in baseline to end of study. To be assessed by standard criteria based on bone marrow examination
Time Frame: Depending on outcomes, will initiate this assessment after 2 years and will continue until completion of study, estimated at 4 years
Population: Relapsed and refractory AML patients who received azacitidine and lenalidomide
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Azacitidine + Lenalidomide + Off Therapy
Number analyzed (Participants) | 37
days | 125 [23 to 308]

4. Secondary Outcome: Toxicity and SAEs Related to Treatment
Description: Change in baseline to end of study. To be measured based on Common Terminology Criteria for Adverse Events (CTCAE) criteria
Time Frame: Will begin assessment with first patient and will continue until completion of study, estimated to be 4 years
Population: Relapsed and refractory AML patients who received azacitidine and lenalidomide -See toxicity data reported for results
Measure: Number; unit: percentage of SAEs related to treatment
Arm/Group | Azacitidine + Lenalidomide + Off Therapy
Number analyzed (Participants) | 37
percentage of SAEs related to treatment | 46

5. Secondary Outcome: Overall Survival
Description: Change in baseline to end of study
Time Frame: Depending on outcomes, will begin assessment at 2 years and will continue until completion of study, estimated to be at four years
Population: Relapsed and refractory AML patients who received azacitidine and lenalidomide
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Azacitidine + Lenalidomide + Off Therapy
Number analyzed (Participants) | 37
days | 166 [35 to 355]

6. Secondary Outcome: Progression-free Survival
Description: Change in baseline to end of study. To be assessed by standard criteria based on bone marrow examination
Time Frame: as for outcome 3
Population: Relapsed and refractory AML patients who received azacitidine and lenalidomide
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Azacitidine + Lenalidomide + Off Therapy
Number analyzed (Participants) | 37
days | 112 [33 to 355]

7. Secondary Outcome: Determine Biomarkers That Predict Response/Toxicity
Description: Change in baseline to end of study. Planned assessments of methylation changes and other biomarkers. Computational biology modeling used to identify biomarkers and predict response.
Time Frame: Three years after initiating study
Population: Relapsed and refractory AML patients who received azacitidine and lenalidomide.
Measure: Number; unit: patients w/response predictor mutations
Arm/Group | Azacitidine + Lenalidomide + Off Therapy
Number analyzed (Participants) | 37
patients w/response predictor mutations | 9

ADVERSE EVENTS:
Arm/Group | Azacitidine + Lenalidomide + Off Therapy
Serious Adverse Events (participants affected / at risk) | 24/37
Other Adverse Events (participants affected / at risk) | 28/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azacitidine + Lenalidomide + Off Therapy (N=37)
Febrile Neutropenia (Blood and lymphatic system disorders) | 11
Clostridium Defficile (Gastrointestinal disorders) | 2
Sepsis (Infections and infestations) | 2
Syncope (Cardiac disorders) | 2
Pneuomonia (Infections and infestations) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Hypertension (Cardiac disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azacitidine + Lenalidomide + Off Therapy (N=37)
Neutropenia (Blood and lymphatic system disorders) | 21
Thrombocytopenia (Blood and lymphatic system disorders) | 12
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 17
Fatigue (General disorders) | 28
Nausea (Gastrointestinal disorders) | 16
Constipation (Gastrointestinal disorders) | 17
Diarrhea (Gastrointestinal disorders) | 21
Anemia (Blood and lymphatic system disorders) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No